CLINICAL TRIAL: NCT03440307
Title: Intervention to Reduce Bisphenol A Exposure in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cal Poly 11/12/2015
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Environmental Exposure

STUDY DESIGN:
Intervention Model Description: Participants randomized to intervention or control.
Who Masked: Outcomes Assessor
Masking Description: Single-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Email Only (Placebo Comparator): Participants received weekly email about health and fitness education. No face-to-face intervention, and not provided any other information about bisphenol exposure.
  Interventions: Behavioral: Email Only
- Face-to-Face Meetings (Experimental): Participants met with a counselor once per week for 3-weeks to reduce bisphenol exposure. Intervention included same weekly email about health and fitness education as Email only group, and a weekly face-to-face meetings to reduce bisphenol exposures from food, cosmetics, and packaged products. Women provided with bisphenol-free cosmetics, hygiene, and glass food/water containers.
  Interventions: Behavioral: Face-to-Face Meetings

INTERVENTIONS:
Behavioral: Face-to-Face Meetings — Participants received health and fitness education, and a face-to-face 3-week intervention to reduce bisphenol exposure.
  Arms: Face-to-Face Meetings
Behavioral: Email Only — Participants received health and fitness education.
  Arms: Email Only

SUMMARY:
The purpose of this study is to determine whether a 3-week intervention reduces urinary Bisphenol A (BPA) in women with obesity

DETAILED DESCRIPTION:
The purpose of this study is reduce BPA exposure in women. The intervention is rooted in social cognitive theory, and is applied to environmental health.

ELIGIBILITY:
Inclusion Criteria:

* BMI >29.9
* Age 18-50 years
* Non-smoking
* English speaking

Exclusion Criteria:

* History of infertility
* Type 2 or Type 1 diabetes
* Cardiovascular disease, or any other metabolic disease/complication
* History of major psychiatric illness, drug abuse, or unsafe dieting practices
* History of bariatric surgery
* Pregnant women or women expecting or trying to become pregnant
* Participating in other studies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women have higher BPA vs. Men
Enrollment: 30 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Urine BPA at 3-weeks | Single urine overnight fasted sample at baseline (date of randomization) and 3-weeks
  Change in urinary BPA measured at baseline and 3-weeks

SECONDARY OUTCOMES:
Change from Baseline Urine BPS and BPF at 3-weeks | Single urine overnight fasted sample at baseline (date of randomization) and 3-weeks
  Change in urinary BPS and BPF measured at baseline and 3-weeks
Change from Baseline Weight at 3-weeks | Overnight fasted weight at baseline (date of randomization) and 3-weeks
  Change in body weight measured at baseline and 3-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Hart, Study Chair — Compliance/Information Officer
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data in this pilot study

REFERENCES:
- [Derived] Hagobian T, Delli-Bovi Z, Mercado A, Bird A, Guy M, Phelan S. Development and feasibility of randomized trial to reduce urinary bisphenols in women with obesity. Pilot Feasibility Stud. 2021 Jan 12;7(1):24. doi: 10.1186/s40814-020-00744-5. PMID 33436090